CLINICAL TRIAL: NCT03803696
Title: Randomized Trial of a Multimodal Sexual Dysfunction Intervention for Hematopoietic Stem Cell Transplant Survivors
Brief Title: Multimodal Sexual Dysfunction Intervention In HCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other); The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-543
Record Dates: First submitted 2019-01-09; First posted 2019-01-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic Stem Cell Transplantation; Hematologic Diseases; Sexual Dysfunction
Keywords: Hematopoietic Stem Cell Transplantation; Hematologic Diseases; Sexual Dysfunction
MeSH Terms: conditions — Hematologic Diseases; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Standard Care (Active Comparator): * Baseline data collection, registration and randomization
  * Inform primary transplant clinician of sexual dysfunction causing distress
  * Receive American Cancer Society sexual educational material
  Interventions: Behavioral: Enhanced Standard Care
- Multimodal Intervention to Address Sexual Dysfunction (Active Comparator): * Baseline data collection, registration and randomization
  * 3 Monthly visits with trained study nurse practitioners
    * Referral to specialist if
    * Psychological etiology
    * Sexual Trauma
    * Relationship Discord
    * Concern for Malignancy or anatomic scarring requiring surgery
  Interventions: Behavioral: Multimodal Intervention to Address Sexual Dysfunction

INTERVENTIONS:
Behavioral: Enhanced Standard Care — * Baseline data collection, registration and randomization
  * Inform primary transplant clinician of sexual dysfunction causing distress
  * Receive American Cancer Society sexual educational material
  Arms: Enhanced Standard Care
Behavioral: Multimodal Intervention to Address Sexual Dysfunction — Baseline data collection, registration and randomization
  - 3 Monthly visits with trained study nurse practitioners
  * Referral to specialist if
  * Psychological etiology
  * Sexual Trauma
  * Relationship Discord
  * Concern for Malignancy or anatomic scarring requiring surgery
  Arms: Multimodal Intervention to Address Sexual Dysfunction

SUMMARY:
This research study is evaluating the impact of an intervention to improve sexual function in stem cell transplant survivors on participants' sexual function, quality of life, and mood.

It is expected that about 120 people who have undergone a stem cell transplant will take part in this research study.

DETAILED DESCRIPTION:
Frequently survivors of stem cell transplantation report significant problems with their sexual function that impacts their quality of life, mood, and their intimacy and relationship with their partners. These issues can be very distressing to patients and their loved ones. The Investigators want to know if the introduction of an intervention focused on improving sexual function may improve a participant's overall care and quality of life.

The main purpose of this study is to compare two types of care - the study intervention versus enhanced standard care which includes receiving an educational handout about sexual dysfunction. The main goal is to assess if the intervention will improve participant's sexual function, quality of life, and mood.

The intervention includes a comprehensive assessment by a transplant clinician (a transplant physician or nurse practitioner) who is trained in sexual dysfunction assessment to explore the reasons for sexual dysfunction and focus on ways to improve symptoms.

-- If the transplant clinician feels additional help is needed by a sexual health expert, the participant will be referred to the sexual health clinic. In the sexual health clinic, the participant will be evaluated by an expert physician who will also focus on strategies to improve sexual function.

The study will use a series of questionnaires to measure sexual function, quality of life, physical symptoms, and mood. Study questionnaires will be completed in the clinic or remotely with assistance provided as needed.

.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) with hematologic malignancy who underwent autologous or allogeneic HCT ≥ three months prior to study enrollment.
* Positive screen for sexual dysfunction that is causing distress based on the National Comprehensive Cancer Network (NCCN) survivorship guidelines
* Ability to read and respond to questions in English or to complete questionnaires with assistance from an interpreter.

Exclusion Criteria:

* Patients with relapsed disease requiring treatment
* Patients with a planned second transplant
* Patients > 5 years from their HCT
* Patients with psychiatric or cognitive conditions which the treating clinicians believes prohibits compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare Patient Global Satisfaction with Sex | 3 Months
  compare patients' global satisfaction with sex using PROMIS Sexual Function and Satisfaction Measure (global satisfaction domain) at three months between the study groups using linear regression controlling for baseline values (as necessary for any imbalances in baseline variables

SECONDARY OUTCOMES:
Compare Patient reported interest in sexual activity | 3 Months
  PROMIS Sexual Function and Satisfaction Measure Interest in sexual activity domain)
Compare Patient global satisfaction with sex longitudinally | up to 6 months
  compare PROMIS Sexual function and Satisfaction Measure - global satisfaction with sex domain) longitudinally between study groups
Compare Patient reported interest in sexual activity longitudinally | up to 6 months
  compare PROMIS Sexual Function and Satisfaction Measure Interest in sexual activity domain) longitudinally between study groups
Compare patient-reported orgasm | 3 Months
  Compare PROMIS Sexual Function and Satisfaction Measure - Orgasm domain
Compare patient-reported orgasm longitudinally | up to 6 months
  Compare PROMIS Sexual Function and Satisfaction Measure - Orgasm domain) longitudinally between the study groups
For males: compare patient-reported erectile function | 3 Months
  PROMIS Sexual Function and Satisfaction Measure - Erectile function domain
For males: compare patient-reported erectile function longitudinally | up to 6 months
  Compare PROMIS Sexual Function and Satisfaction Measure - Erectile function domain longitudinally between the two groups
For females: compare patient-reported vaginal lubrication | 3 Months
  compare (PROMIS Sexual Function and Satisfaction Measure - lubrication domain)
For females: compare patient-reported vaginal lubrication longitudinally | up to 6 months
  compare (PROMIS Sexual Function and Satisfaction Measure - lubrication domain) longitudinally between the two study groups
For females: compare patient-reported vaginal comfort | 3 months
  compare (PROMIS Sexual Function and Satisfaction Measure - vaginal comfort domain
For females: compare patient-reported vaginal comfort longitudinally | up to 6 months
  compare (PROMIS Sexual Function and Satisfaction Measure - vaginal comfort domain) longitudinally between the two study groups
Compare Patient Reported Quality of Life | 3 Months
  Compare patient-reported QOL using the Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT)
Compare Patient Reported Quality of Life longitudinally | up to 6 months
  Compare patient-reported QOL using the Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT) longitudinally between the two groups
Compare Patient Reported Anxiety Symptoms | 3 Months
  Compare patient reported anxiety symptoms using the Hospital Anxiety and Depression Scale (HADS- anxiety subscale). Subscale ranges from 0-21 with higher score indicating higher anxiety symptoms
Compare Patient Reported Anxiety Symptoms Longitudinally | up to 6 months
  Compare patient reported anxiety symptoms using the Hospital Anxiety and Depression Scale (HADS- anxiety subscale) longitudinally between the two study groups. Subscale ranges from 0-21 with higher score indicating higher anxiety symptoms
Compare Patient Reported Depression Symptoms | 3 Months
  Compare Patient Reported Depression Symptoms using the Hospital Anxiety and Depression Scale (HADS - depression subscale). Subscale ranges from 0-21 with higher score indicating higher depression symptoms
Compare Patient Reported Depression Symptoms Longitudinally | up to 6 Months
  Compare Patient Reported Depression Symptoms using the Hospital Anxiety and Depression Scale (HADS - depression subscale) longitudinally between the two study groups. Subscale ranges from 0-21 with higher score indicating higher depression symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawhri, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Requests may be directed to:MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] El-Jawahri A, Traeger L, Reese JB, Dizon D, Bober SL, Greer JA, Vanderklish J, Horick N, Ufere N, Reynolds MJ, Rice J, Clay M, Newcomb R, DeFilipp Z, Chen YB, Temel JS. A multimodal sexual dysfunction intervention versus enhanced usual care for survivors of haematopoietic stem-cell transplantation: a single-centre, open-label, randomised clinical trial. Lancet Haematol. 2025 Aug;12(8):e611-e620. doi: 10.1016/S2352-3026(25)00160-7. PMID 40769685